CLINICAL TRIAL: NCT01755598
Title: Efficacy of GSK Biologicals' Candidate Tuberculosis (TB) Vaccine GSK 692342 Against TB Disease, in Adults Living in a TB Endemic Region
Brief Title: Study to Evaluate the Efficacy of GlaxoSmithKline (GSK) Biologicals' Candidate Tuberculosis (TB) Vaccine in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Aeras (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 115616
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Results first posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Tuberculosis; Tuberculosis Vaccines
Keywords: Positive Interferon-γ release assay; Efficacy; Adults; Tuberculosis vaccine; Endemic region
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M72AS01 Group (Experimental): Subjects, between, and including, 18 and 50 years of age, who received 2 doses of M72/AS01E according to random assignment, one month apart (Day 0 and Day 30) by intramuscular injection in the deltoid region of the arm.
  Interventions: Biological: GSK Biologicals' investigational TB vaccine (GSK692342)
- Control group (Placebo Comparator): Subjects, between, and including,18 and 50 years of age, who received 2 doses of Placebo according to random assignment, one month apart (Day 0 and Day 30) by intramuscular injection in the deltoid region of the arm.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: GSK Biologicals' investigational TB vaccine (GSK692342) — 2 doses administered intramuscularly in the deltoid region of the arm.
  Arms: M72AS01 Group
Biological: Placebo — 2 doses administered intramuscularly in the deltoid region of the arm.
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate the protective efficacy of two doses of GSK Biologicals' candidate TB vaccine against pulmonary TB, as compared to placebo. The efficacy will be evaluated in adults living in TB endemic countries and aged 18 - 50 years because pulmonary TB occurs frequently in these countries and age range. In addition, the safety and immunogenicity of the candidate tuberculosis vaccine will be evaluated in a subset of volunteers.

DETAILED DESCRIPTION:
Case Definitions:

• First case definition: A subject with clinical suspicion of pulmonary TB disease, with MTB complex identified from a sputum specimen, taken before initiation of TB treatment, by Xpert MTB/RIF and/or microbiological culture and confirmed HIV-negative at the time of TB diagnosis.

• Second case definition: A subject with clinical suspicion of pulmonary TB disease, with MTB complex identified from a sputum specimen, taken before initiation of TB treatment, by Xpert MTB/RIF and confirmed HIV-negative at the time of TB diagnosis.

• Third case definition: A subject with clinical suspicion of pulmonary TB disease, with MTB complex identified from a sputum specimen, taken up to four weeks after initiation of TB treatment, by Xpert MTB/RIF and/or microbiological culture and confirmed HIV-negative at the time of TB diagnosis.

• Fourth case definition: A subject with clinical suspicion of pulmonary TB disease, with MTB complex identified from a sputum specimen, taken up to four weeks after initiation of TB treatment, by Xpert MTB/RIF and/or microbiological culture.

• Fifth case definition: A subject for whom a clinician has diagnosed TB disease and has decided to treat the patient with TB treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or female between, and including, 18 and 50 years of age at the time of obtaining informed consent.
* Written (or thumb printed and witnessed) informed consent obtained from the subject.
* Baseline positive IGRA test result.
* Baseline negative HIV screen.
* Baseline negative clinical screening questionnaire and negative sputum sample for Pulmonary TB disease.
* Healthy subjects or those with chronic well-controlled disease as established by medical history and clinical examination.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 25 days prior to vaccination, and
  * has a negative pregnancy test on the day of screening and the day of first vaccination, and
  * has agreed to continue adequate contraception during the entire vaccination period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Current TB disease or history of TB disease and/or treatment for TB.
* Use of any investigational or non-registered product other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before and ending 30 days after each dose of vaccine.
* History of previous administration of experimental Mtb vaccines.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose. Inhaled and topical steroids are allowed.
* Any condition or illness or medication, which in the opinion of the Investigator might interfere with the evaluation of the safety or immunogenicity of the vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Planned participation or participation in another experimental protocol during the study.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* History of medically confirmed autoimmune disease.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions during the vaccination period and/or before 2 months after completion of the vaccination series.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3575 (Actual)
Dates: Start 2014-08-19 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (8):
- GSK Investigational Site, Kisumu, Kenya
- South Africa (6):
  - GSK Investigational Site, Pretoria, Gauteng
  - GSK Investigational Site, Soweto, Gauteng
  - GSK Investigational Site, Klerksdorp, North West
  - GSK Investigational Site, Western Cape, Western Province
  - GSK Investigational Site, Worcester, Western Province
  - GSK Investigational Site, Cape Town
- GSK Investigational Site, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20104

REFERENCES:
- [Derived] Tait DR, Hatherill M, Van Der Meeren O, Ginsberg AM, Van Brakel E, Salaun B, Scriba TJ, Akite EJ, Ayles HM, Bollaerts A, Demoitie MA, Diacon A, Evans TG, Gillard P, Hellstrom E, Innes JC, Lempicki M, Malahleha M, Martinson N, Mesia Vela D, Muyoyeta M, Nduba V, Pascal TG, Tameris M, Thienemann F, Wilkinson RJ, Roman F. Final Analysis of a Trial of M72/AS01E Vaccine to Prevent Tuberculosis. N Engl J Med. 2019 Dec 19;381(25):2429-2439. doi: 10.1056/NEJMoa1909953. Epub 2019 Oct 29. PMID 31661198
- [Derived] Van Der Meeren O, Hatherill M, Nduba V, Wilkinson RJ, Muyoyeta M, Van Brakel E, Ayles HM, Henostroza G, Thienemann F, Scriba TJ, Diacon A, Blatner GL, Demoitie MA, Tameris M, Malahleha M, Innes JC, Hellstrom E, Martinson N, Singh T, Akite EJ, Khatoon Azam A, Bollaerts A, Ginsberg AM, Evans TG, Gillard P, Tait DR. Phase 2b Controlled Trial of M72/AS01E Vaccine to Prevent Tuberculosis. N Engl J Med. 2018 Oct 25;379(17):1621-1634. doi: 10.1056/NEJMoa1803484. Epub 2018 Sep 25. PMID 30280651

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 3575 subjects enrolled in the study, 2 subjects did not get any vaccination and therefore were not included in any analysis.
Period: Overall Study
Arm/Group | M72AS01 Group | Control Group
Started | 1786 | 1787
Completed | 1521 | 1504
Not Completed | 265 | 283
Not completed — Other | 109 | 109
Not completed — Lost to Follow-up | 32 | 43
Not completed — Migrated/moved from study area | 76 | 65
Not completed — Withdrawal by Subject | 22 | 31
Not completed — Protocol Violation | 7 | 7
Not completed — Adverse Event | 19 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | M72AS01 Group | Control Group | Total
Number analyzed (Participants) | 1786 | 1787 | 3573
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.9 (8.3) | 28.9 (8.3) | 28.9 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 763 | 766 | 1529
  Male | 1023 | 1021 | 2044
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Heritage / African American | 1346 | 1329 | 2675
  Other, Not Specified | 440 | 458 | 898

OUTCOME MEASURES:

1. Primary Outcome: Incident Rates of Definite Pulmonary Tuberculosis (TB) Disease, Not Associated With HIV-infection, Meeting the Case Definition 1
Description: The incidence rate of definite pulmonary TB disease (or 100 Person-years rate) was calculated as the number of subjects reporting at least one case (n) in a group, over the sum of follow-up period expressed in years (T) in the same group, and multiplied by 100. Case definition 1 = subject with clinical suspicion of pulmonary TB disease*, with Mycobacterium tuberculosis (Mtb) complex identified from sputum specimen, taken before initiation of TB treatment, by Xpert MTB/RIF (Nucleic Acid Amplification Test to detect Mtb complex and resistance to rifampicin in sputum samples) and/or microbiological culture and confirmed Human Immunodeficiency Virus (HIV)-negative at the time of TB diagnosis. *Clinical suspicion of pulmonary TB defined as subject presenting with 1 or more of the following symptoms: unexplained cough > 2 weeks, unexplained fever > 1 week, night sweats, unintentional weight loss, pleuritic chest pains, haemoptysis, fatigue or shortness of breath on exertion.
Time Frame: From Day 60 (i.e one month after Dose 2) up to Year 3: follow-up period for cases ends at the first occurrence of an event. For the non-cases: follow-up period ends at the date of the Month 36 visit or last contact date whichever comes first
Population: Analysis was performed on the According-to-Protocol cohort for efficacy which included all subjects who received all vaccinations according to protocol procedures within specified intervals that contributed time at risk in the follow-up period starting one month post dose 2 (Day 60).
Measure: Number (90% Confidence Interval); unit: cases per 100 person-years
Arm/Group | M72AS01 Group | Control Group
Number analyzed (Participants) | 1626 | 1663
cases per 100 person-years | 0.3 [0.2 to 0.5] | 0.6 [0.4 to 0.8]
Statistical Analysis 1: Comparison: M72AS01 Group vs Control Group; To evaluate the protective efficacy of two doses of the M72/AS01E candidate vaccine against Definite pulmonary TB disease not associated with HIV-infection, meeting the case definition 1, as compared to placebo; Test type: Other — Vaccine efficacy (VE) has been estimated from a Cox proportional hazard regression model (VE=1-hazard ratio) and 90% confidence intervals (CIs) and Wald p-value has been derived. The lower limit of the 90% two-sided CI for the VE against first occurrence of Definite pulmonary TB disease not associated with HIV-infection, meeting the case definition 1, is to be above 0%; p = 0.0430, Regression, Cox; Vaccine efficacy rate = 49.7, 90% CI 2-sided [12.1 to 71.2]

2. Secondary Outcome: Incident Rates of Definite Xpert MTB/Rif Positive Pulmonary TB Disease, Not Associated With HIV-infection, Meeting the Case Definition 2
Description: The incidence rate of definite Xpert MTB/Rif positive pulmonary TB disease, expressed in terms of 100 Person-years rate, was calculated as the number of subjects reporting at least one case (n) in a group over the sum of follow-up period expressed in years (T) in the same group, and multiplied by 100. Case definition 2 = a subject with clinical suspicion* of pulmonary TB disease, with Mtb complex identified from a sputum specimen, taken before initiation of TB treatment, by Xpert MTB/RIF and confirmed HIV-negative at the time of TB diagnosis. *Clinical suspicion of pulmonary TB was defined as a subject presenting with one or more of the following symptoms: unexplained cough > 2 weeks, unexplained fever > 1 week, night sweats, unintentional weight loss, pleuritic chest pains, haemoptysis, fatigue or shortness of breath on exertion.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: cases per 100 person-years
Arm/Group | M72AS01 Group | Control Group
Number analyzed (Participants) | 1626 | 1663
cases per 100 person-years | 0.181 [0.101 to 0.323] | 0.470 [0.328 to 0.673]
Statistical Analysis 1: Comparison: M72AS01 Group vs Control Group; To evaluate the protective efficacy of two doses of the M72/AS01E candidate vaccine against Definite Xpert MTB/Rif positive pulmonary TB disease not associated with HIV-infection, meeting the case definition 2, as compared to placebo; Test type: Other — Vaccine efficacy (VE) has been estimated from a Cox proportional hazard regression model (VE=1-hazard ratio) and 90% confidence intervals (CIs) and Wald p-value has been derived. If the primary objective is met, this secondary objective is to be analysed using the following success criterion: The lower limit of the 90% two-sided CI for the VE against first occurrence of Definite pulmonary TB disease not associated with HIV infection, meeting the case definition 2, is to be above 0%; p = 0.0210, Regression, Cox; Vaccine efficacy rate = 61.670, 90% CI 2-sided [24.084 to 80.647]

3. Secondary Outcome: Incident Rates of Definite Pulmonary TB Disease, Not Associated With HIV-infection Meeting the Case Definition 3
Description: The incidence rate of definite pulmonary TB disease (or 100 Person-years rate) was calculated as the number of subjects reporting at least one case (n) in a group, over the sum of follow-up period expressed in years (T) in the same group, and multiplied by 100. Case definition 3 = a subject with clinical suspicion* of pulmonary TB disease, with Mtb complex identified from a sputum specimen, taken up to four weeks after initiation of TB treatment, by Xpert MTB/RIF and/or microbiological culture and confirmed HIV-negative at the time of TB diagnosis.*Clinical suspicion of pulmonary TB was defined as a subject presenting with one or more of the following symptoms: unexplained cough > 2 weeks, unexplained fever > 1 week, night sweats, unintentional weight loss, pleuritic chest pains, haemoptysis, fatigue or shortness of breath on exertion.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: cases per 100 person-years
Arm/Group | M72AS01 Group | Control Group
Number analyzed (Participants) | 1626 | 1663
cases per 100 person-years | 0.429 [0.294 to 0.626] | 0.672 [0.498 to 0.908]

4. Secondary Outcome: Incident Rates of Microbiological Pulmonary TB Disease, Meeting the Case Definition 4
Description: The incidence rate of Microbiological pulmonary TB disease (or 100 Person-years rate) was calculated as the number of subjects reporting at least one case (n) in a group, over the sum of follow-up period expressed in years (T) in the same group, and multiplied by 100. Case definition 4 = a subject with clinical suspicion* of pulmonary TB disease, with Mtb complex identified from a sputum specimen, taken up to four weeks after initiation of TB treatment, by Xpert MTB/RIF and/or microbiological culture.*Clinical suspicion of pulmonary TB was defined as a subject presenting with one or more of the following symptoms: unexplained cough > 2 weeks, unexplained fever > 1 week, night sweats, unintentional weight loss, pleuritic chest pains, haemoptysis, fatigue or shortness of breath on exertion.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: cases per 100 person-years
Arm/Group | M72AS01 Group | Control Group
Number analyzed (Participants) | 1626 | 1663
cases per 100 person-years | 0.429 [0.294 to 0.626] | 0.717 [0.536 to 0.959]

5. Secondary Outcome: Incidence Rates of Clinical TB Disease, Meeting the Case Definition 5
Description: The incidence rate of Clinical TB disease (or 100 Person-years rate) was calculated as the number of subjects reporting at least one case (n) in a group, over the sum of follow-up period expressed in years (T) in the same group, and multiplied by 100. Case definition 5 = a subject for whom a clinician has diagnosed TB disease and has decided to treat the patient with TB treatment.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: cases per 100 person-years
Arm/Group | M72AS01 Group | Control Group
Number analyzed (Participants) | 1626 | 1663
cases per 100 person-years | 0.586 [0.425 to 0.810] | 0.850 [0.651 to 1.109]

6. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs).
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Day 0 up to Year 3 (during the entire study period)
Population: Analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects with at least one dose administered.
Measure: Count of Participants; unit: Participants
Arm/Group | M72AS01 Group | Control Group
Number analyzed (Participants) | 1786 | 1787
Participants | 51 | 62

7. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs).
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 30-day follow-up period following vaccination, across doses (i.e. day of vaccination and 29 subsequent days after each vaccine dose)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | M72AS01 Group | Control Group
Number analyzed (Participants) | 1786 | 1787
Participants | 1207 | 816

8. Secondary Outcome: Number of Subjects With Any Solicited Local AEs in the Safety and Immune Sub-cohort
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Any redness/swelling symptom was scored as injection site redness/swelling with a diameter equal or larger than (≥) 20 millimeters (mm).
Time Frame: During the 7-day follow-up period (i.e. day of vaccination and 6 subsequent days) after each vaccine dose
Population: Analysis was performed on the "safety and immunogenicity" sub-cohort (i.e. about 150 subjects enrolled in each group and from 2 of the 3 countries [the third country study start was delayed as awaiting regulatory approval]) which included subjects with at least 1 vaccination dose documented.
Measure: Count of Participants; unit: Participants
Arm/Group | M72AS01 Group | Control Group
Number analyzed (Participants) | 148 | 151
Participants
  Any Pain after Dose 1 | 111 | 48
  Any Redness after Dose 1 | 12 | 0
  Any Swelling after Dose 1 | 25 | 1
  Any Pain after Dose 2: number analyzed (Participants) | 130 | 141
  Any Pain after Dose 2 | 86 | 22
  Any Redness after Dose 2: number analyzed (Participants) | 130 | 141
  Any Redness after Dose 2 | 5 | 2
  Any Swelling after Dose 2: number analyzed (Participants) | 130 | 141
  Any Swelling after Dose 2 | 12 | 2

9. Secondary Outcome: Number of Subjects With Any Solicited General AEs in the Safety and Immune Sub-cohort
Description: Assessed solicited general symptoms were fatigue, fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)], respiratory symptoms (including cough, blood in sputum, purulent sputum, shortness of breath or difficulties breathing, chest wall pain) headache, malaise and myalgia. Any = occurrence of the symptom regardless of intensity grade and relation to vaccination.
Time Frame: During the 7-day follow-up period (i.e.: day of vaccination and 6 subsequent days) after each vaccine dose
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | M72AS01 Group | Control Group
Number analyzed (Participants) | 148 | 151
Participants
  Any Fatigue after Dose 1 | 91 | 63
  Any Headache after Dose 1 | 81 | 60
  Any Malaise after Dose 1 | 68 | 29
  Any Myalgia after Dose 1 | 75 | 34
  Any Respiratory symptoms after Dose 1 | 23 | 13
  Any Fever after Dose 1 | 33 | 16
  Any Fatigue after Dose 2: number analyzed (Participants) | 130 | 141
  Any Fatigue after Dose 2 | 70 | 31
  Any Headache after Dose 2: number analyzed (Participants) | 130 | 141
  Any Headache after Dose 2 | 75 | 39
  Any Malaise after Dose 2: number analyzed (Participants) | 130 | 141
  Any Malaise after Dose 2 | 57 | 21
  Any Myalgia after Dose 2: number analyzed (Participants) | 130 | 141
  Any Myalgia after Dose 2 | 55 | 21
  Any Respiratory symptoms after Dose 2: number analyzed (Participants) | 130 | 141
  Any Respiratory symptoms after Dose 2 | 14 | 5
  Any Fever after Dose 2: number analyzed (Participants) | 130 | 141
  Any Fever after Dose 2 | 37 | 10

10. Secondary Outcome: Number of Subjects With Any Potential Immune-mediated Diseases (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: From Day 0 to 6 months post-dose 2 (i.e. at Month 7)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | M72AS01 Group | Control Group
Number analyzed (Participants) | 1786 | 1787
Participants | 2 | 6

11. Secondary Outcome: Number of Subjects With Grade Equal or Greater Than 2 of Severity for Haematological and Biochemichal Abnormal Laboratory Values in the Safety and Immune Sub-cohort
Description: Abnormal laboratory values include haematological abnormalities (haemoglobin level, white blood cells and platelets) and biochemical abnormalities (alanine aminotransferase, aspartate aminotransferase and creatinine). Grading was defined based on the Food and Drug Administration [FDA], 2007. Guidance for Industry, Toxicity Grading Scale for Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials. Alanine Aminotransferase = ALA; Aspartate Aminotransferase = ASP; Creatinine = CREA; Hemoglobin (Change from baseline) = HEM (baseline); Hemoglobin (decrease) = HEM (decrease); Leukocytes (White Blood Cells) (Decrease) = WBC (decrease); Leukocytes (White Blood Cells) (Increase) = WBC (increase); Platelets = PLA; Total Bilirubin = BIL.
Time Frame: Days 0, 7, 30 and 37
Population: Analysis was performed on the "safety and immunogenicity" sub-cohort (i.e. about 150 subjects enrolled in each group and from 2 of the 3 countries [the third country study start was delayed as awaiting regulatory approval]) which included subjects with at least 1 laboratory value documented.
Measure: Count of Participants; unit: Participants
Arm/Group | M72AS01 Group | Control Group
Number analyzed (Participants) | 149 | 151
Participants
  Grade 2 ALA at Day 0 | 0 | 0
  Grade 3 ALA at Day 0 | 0 | 0
  Grade 4 ALA at Day 0 | 0 | 0
  Grade 2 ALA at Day 7: number analyzed (Participants) | 149 | 146
  Grade 2 ALA at Day 7 | 0 | 0
  Grade 3 ALA at Day 7: number analyzed (Participants) | 149 | 146
  Grade 3 ALA at Day 7 | 0 | 0
  Grade 4 ALA at Day 7: number analyzed (Participants) | 149 | 146
  Grade 4 ALA at Day 7 | 0 | 0
  Grade 2 ALA at Day 30: number analyzed (Participants) | 139 | 151
  Grade 2 ALA at Day 30 | 0 | 0
  Grade 3 ALA at Day 30: number analyzed (Participants) | 139 | 151
  Grade 3 ALA at Day 30 | 0 | 0
  Grade 4 ALA at Day 30: number analyzed (Participants) | 139 | 151
  Grade 4 ALA at Day 30 | 0 | 0
  Grade 2 ALA at Day 37: number analyzed (Participants) | 122 | 136
  Grade 2 ALA at Day 37 | 0 | 0
  Grade 3 ALA at Day 37: number analyzed (Participants) | 122 | 136
  Grade 3 ALA at Day 37 | 0 | 0
  Grade 4 ALA at Day 37: number analyzed (Participants) | 122 | 136
  Grade 4 ALA at Day 37 | 0 | 0
  Grade 2 ASP at Day 0 | 1 | 0
  Grade 3 ASP at Day 0 | 0 | 0
  Grade 4 ASP at Day 0 | 0 | 0
  Grade 2 ASP at Day 7: number analyzed (Participants) | 149 | 146
  Grade 2 ASP at Day 7 | 1 | 0
  Grade 3 ASP at Day 7: number analyzed (Participants) | 149 | 146
  Grade 3 ASP at Day 7 | 0 | 0
  Grade 4 ASP at Day 7: number analyzed (Participants) | 149 | 146
  Grade 4 ASP at Day 7 | 0 | 0
  Grade 2 ASP at Day 30: number analyzed (Participants) | 139 | 151
  Grade 2 ASP at Day 30 | 0 | 0
  Grade 3 ASP at Day 30: number analyzed (Participants) | 139 | 151
  Grade 3 ASP at Day 30 | 0 | 0
  Grade 4 ASP at Day 30: number analyzed (Participants) | 139 | 151
  Grade 4 ASP at Day 30 | 0 | 0
  Grade 2 ASP at Day 37: number analyzed (Participants) | 122 | 136
  Grade 2 ASP at Day 37 | 0 | 0
  Grade 3 ASP at Day 37: number analyzed (Participants) | 122 | 136
  Grade 3 ASP at Day 37 | 1 | 0
  Grade 4 ASP at Day 37: number analyzed (Participants) | 122 | 136
  Grade 4 ASP at Day 37 | 0 | 0
  Grade 2 CREA at Day 0 | 0 | 0
  Grade 3 CREA at Day 0 | 0 | 0
  Grade 4 CREA at Day 0 | 0 | 0
  Grade 2 CREA at Day 7: number analyzed (Participants) | 149 | 146
  Grade 2 CREA at Day 7 | 0 | 0
  Grade 3 CREA at Day 7: number analyzed (Participants) | 149 | 146
  Grade 3 CREA at Day 7 | 0 | 0
  Grade 4 CREA at Day 7: number analyzed (Participants) | 149 | 146
  Grade 4 CREA at Day 7 | 0 | 0
  Grade 2 CREA at Day 30: number analyzed (Participants) | 139 | 151
  Grade 2 CREA at Day 30 | 0 | 0
  Grade 3 CREA at Day 30: number analyzed (Participants) | 139 | 151
  Grade 3 CREA at Day 30 | 0 | 0
  Grade 4 CREA at Day 30: number analyzed (Participants) | 139 | 151
  Grade 4 CREA at Day 30 | 0 | 0
  Grade 2 CREA at Day 37: number analyzed (Participants) | 122 | 136
  Grade 2 CREA at Day 37 | 0 | 0
  Grade 3 CREA at Day 37: number analyzed (Participants) | 122 | 136
  Grade 3 CREA at Day 37 | 0 | 0
  Grade 4 CREA at Day 37: number analyzed (Participants) | 122 | 136
  Grade 4 CREA at Day 37 | 0 | 0
  Grade 2 HEM (baseline) at Day 0 | 0 | 0
  Grade 3 HEM (baseline) at Day 0 | 0 | 0
  Grade 4 HEM (baseline) at Day 0 | 0 | 0
  Grade 2 HEM (baseline) at Day 7: number analyzed (Participants) | 149 | 146
  Grade 2 HEM (baseline) at Day 7 | 1 | 5
  Grade 3 HEM (baseline) at Day 7: number analyzed (Participants) | 149 | 146
  Grade 3 HEM (baseline) at Day 7 | 0 | 0
  Grade 4 HEM (baseline) at Day 7: number analyzed (Participants) | 149 | 146
  Grade 4 HEM (baseline) at Day 7 | 0 | 0
  Grade 2 HEM (baseline) at Day 30: number analyzed (Participants) | 139 | 151
  Grade 2 HEM (baseline) at Day 30 | 2 | 2
  Grade 3 HEM (baseline) at Day 30: number analyzed (Participants) | 139 | 151
  Grade 3 HEM (baseline) at Day 30 | 0 | 0
  Grade 4 HEM (baseline) at Day 30: number analyzed (Participants) | 139 | 151
  Grade 4 HEM (baseline) at Day 30 | 0 | 0
  Grade 2 HEM (baseline) at Day 37: number analyzed (Participants) | 122 | 136
  Grade 2 HEM (baseline) at Day 37 | 2 | 0
  Grade 3 HEM (baseline) at Day 37: number analyzed (Participants) | 122 | 136
  Grade 3 HEM (baseline) at Day 37 | 1 | 0
  Grade 4 HEM (baseline) at Day 37: number analyzed (Participants) | 122 | 136
  Grade 4 HEM (baseline) at Day 37 | 0 | 0
  Grade 2 HEM (decrease) at Day 0 | 5 | 5
  Grade 3 HEM (decrease) at Day 0 | 2 | 1
  Grade 4 HEM (decrease) at Day 0 | 1 | 0
  Grade 2 HEM (decrease) at Day 7: number analyzed (Participants) | 149 | 146
  Grade 2 HEM (decrease) at Day 7 | 10 | 5
  Grade 3 HEM (decrease) at Day 7: number analyzed (Participants) | 149 | 146
  Grade 3 HEM (decrease) at Day 7 | 2 | 2
  Grade 4 HEM (decrease) at Day 7: number analyzed (Participants) | 149 | 146
  Grade 4 HEM (decrease) at Day 7 | 0 | 0
  Grade 2 HEM (decrease) at Day 30: number analyzed (Participants) | 139 | 151
  Grade 2 HEM (decrease) at Day 30 | 5 | 4
  Grade 3 HEM (decrease) at Day 30: number analyzed (Participants) | 139 | 151
  Grade 3 HEM (decrease) at Day 30 | 2 | 1
  Grade 4 HEM (decrease) at Day 30: number analyzed (Participants) | 139 | 151
  Grade 4 HEM (decrease) at Day 30 | 0 | 0
  Grade 2 HEM (decrease) at Day 37: number analyzed (Participants) | 122 | 136
  Grade 2 HEM (decrease) at Day 37 | 4 | 4
  Grade 3 HEM (decrease) at Day 37: number analyzed (Participants) | 122 | 136
  Grade 3 HEM (decrease) at Day 37 | 1 | 0
  Grade 4 HEM (decrease) at Day 37: number analyzed (Participants) | 122 | 136
  Grade 4 HEM (decrease) at Day 37 | 0 | 0
  Grade 2 WBC (decrease) at Day 0 | 0 | 0
  Grade 3 WBC (decrease) at Day 0 | 0 | 0
  Grade 4 WBC (decrease) at Day 0 | 0 | 0
  Grade 2 WBC (decrease) at Day 7: number analyzed (Participants) | 149 | 146
  Grade 2 WBC (decrease) at Day 7 | 0 | 0
  Grade 3 WBC (decrease) at Day 7: number analyzed (Participants) | 149 | 146
  Grade 3 WBC (decrease) at Day 7 | 0 | 0
  Grade 4 WBC (decrease) at Day 7: number analyzed (Participants) | 149 | 146
  Grade 4 WBC (decrease) at Day 7 | 0 | 0
  Grade 2 WBC (decrease) at Day 30: number analyzed (Participants) | 139 | 151
  Grade 2 WBC (decrease) at Day 30 | 0 | 0
  Grade 3 WBC (decrease) at Day 30: number analyzed (Participants) | 139 | 151
  Grade 3 WBC (decrease) at Day 30 | 0 | 0
  Grade 4 WBC (decrease) at Day 30: number analyzed (Participants) | 139 | 151
  Grade 4 WBC (decrease) at Day 30 | 0 | 0
  Grade 2 WBC (decrease) at Day 37: number analyzed (Participants) | 122 | 136
  Grade 2 WBC (decrease) at Day 37 | 0 | 0
  Grade 3 WBC (decrease) at Day 37: number analyzed (Participants) | 122 | 136
  Grade 3 WBC (decrease) at Day 37 | 0 | 0
  Grade 4 WBC (decrease) at Day 37: number analyzed (Participants) | 122 | 136
  Grade 4 WBC (decrease) at Day 37 | 0 | 0
  Grade 2 WBC (increase) at Day 0 | 0 | 0
  Grade 3 WBC (increase) at Day 0 | 0 | 0
  Grade 4 WBC (increase) at Day 0 | 0 | 0
  Grade 2 WBC (increase) at Day 7: number analyzed (Participants) | 149 | 146
  Grade 2 WBC (increase) at Day 7 | 0 | 0
  Grade 3 WBC (increase) at Day 7: number analyzed (Participants) | 149 | 146
  Grade 3 WBC (increase) at Day 7 | 0 | 0
  Grade 4 WBC (increase) at Day 7: number analyzed (Participants) | 149 | 146
  Grade 4 WBC (increase) at Day 7 | 0 | 0
  Grade 2 WBC (increase) at Day 30: number analyzed (Participants) | 139 | 151
  Grade 2 WBC (increase) at Day 30 | 0 | 0
  Grade 3 WBC (increase) at Day 30: number analyzed (Participants) | 139 | 151
  Grade 3 WBC (increase) at Day 30 | 0 | 0
  Grade 4 WBC (increase) at Day 30: number analyzed (Participants) | 139 | 151
  Grade 4 WBC (increase) at Day 30 | 0 | 0
  Grade 2 WBC (increase) at Day 37: number analyzed (Participants) | 122 | 136
  Grade 2 WBC (increase) at Day 37 | 0 | 0
  Grade 3 WBC (increase) at Day 37: number analyzed (Participants) | 122 | 136
  Grade 3 WBC (increase) at Day 37 | 0 | 0
  Grade 4 WBC (increase) at Day 37: number analyzed (Participants) | 122 | 136
  Grade 4 WBC (increase) at Day 37 | 0 | 0
  Grade 2 PLA at Day 0 | 3 | 2
  Grade 3 PLA at Day 0 | 4 | 0
  Grade 4 PLA at Day 0 | 0 | 0
  Grade 2 PLA at Day 7: number analyzed (Participants) | 149 | 146
  Grade 2 PLA at Day 7 | 0 | 1
  Grade 3 PLA at Day 7: number analyzed (Participants) | 149 | 146
  Grade 3 PLA at Day 7 | 3 | 0
  Grade 4 PLA at Day 7: number analyzed (Participants) | 149 | 146
  Grade 4 PLA at Day 7 | 0 | 0
  Grade 2 PLA at Day 30: number analyzed (Participants) | 139 | 151
  Grade 2 PLA at Day 30 | 1 | 3
  Grade 3 PLA at Day 30: number analyzed (Participants) | 139 | 151
  Grade 3 PLA at Day 30 | 3 | 1
  Grade 4 PLA at Day 30: number analyzed (Participants) | 139 | 151
  Grade 4 PLA at Day 30 | 0 | 0
  Grade 2 PLA at Day 37: number analyzed (Participants) | 122 | 136
  Grade 2 PLA at Day 37 | 1 | 1
  Grade 3 PLA at Day 37: number analyzed (Participants) | 122 | 136
  Grade 3 PLA at Day 37 | 3 | 0
  Grade 4 PLA at Day 37: number analyzed (Participants) | 122 | 136
  Grade 4 PLA at Day 37 | 0 | 0
  Grade 2 BIL at Day 0 | 1 | 4
  Grade 3 BIL at Day 0 | 0 | 0
  Grade 4 BIL at Day 0 | 0 | 1
  Grade 2 BIL at Day 7: number analyzed (Participants) | 149 | 146
  Grade 2 BIL at Day 7 | 0 | 1
  Grade 3 BIL at Day 7: number analyzed (Participants) | 149 | 146
  Grade 3 BIL at Day 7 | 0 | 1
  Grade 4 BIL at Day 7: number analyzed (Participants) | 149 | 146
  Grade 4 BIL at Day 7 | 0 | 1
  Grade 2 BIL at Day 30: number analyzed (Participants) | 139 | 151
  Grade 2 BIL at Day 30 | 1 | 1
  Grade 3 BIL at Day 30: number analyzed (Participants) | 139 | 151
  Grade 3 BIL at Day 30 | 1 | 1
  Grade 4 BIL at Day 30: number analyzed (Participants) | 139 | 151
  Grade 4 BIL at Day 30 | 3 | 1
  Grade 2 BIL at Day 37: number analyzed (Participants) | 122 | 136
  Grade 2 BIL at Day 37 | 1 | 2
  Grade 3 BIL at Day 37: number analyzed (Participants) | 122 | 136
  Grade 3 BIL at Day 37 | 0 | 0
  Grade 4 BIL at Day 37: number analyzed (Participants) | 122 | 136
  Grade 4 BIL at Day 37 | 0 | 0

12. Secondary Outcome: Desciptive Statistics of the Frequency of M72-specific CD4+ T-cells Expressing Any Combination of Immune Markers in the Safety and Immune Sub-cohort
Description: The frequency of M72-specific CD4 + T-cells per million cells were identified after in vitro stimulation expressing any combination of immune markers ( Interleukin-2 (IL-2), cluster of differentiation 40-ligand (CD40-L), tumor necrosis factor alpha (TNF-) and interferon-gamma (IFN-) after background subtraction for each treatment group.
Time Frame: Prior to dose 1 (Day 0) and post-dose 2 (Day 60, Year 1, Year 2 and Year 3)
Population: Analysis was performed on the "safety and immunogenicity" sub-cohort (i.e. about 150 subjects enrolled in each group and from 2 of the 3 countries [the third country study start was delayed as awaiting regulatory approval]) which included subjects with at least 1 immune result documented.
Measure: Median (Inter-Quartile Range); unit: T cells per million cells
Arm/Group | M72AS01 Group | Control Group
Number analyzed (Participants) | 84 | 84
T cells per million cells
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+) at Day 0: number analyzed (Participants) | 71 | 69
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+) at Day 0 | 1.0 [1.0 to 178.0] | 28.0 [1.0 to 135.0]
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+) at Day 60: number analyzed (Participants) | 51 | 48
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+) at Day 60 | 1.0 [1.0 to 227.0] | 1.0 [1.0 to 86.5]
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+) at Year 1: number analyzed (Participants) | 84 | 79
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+) at Year 1 | 300.5 [66.5 to 831.5] | 53.0 [1.0 to 255.0]
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+) at Year 2: number analyzed (Participants) | 76 | 84
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+) at Year 2 | 1.0 [1.0 to 480.0] | 1.0 [1.0 to 113.5]
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+) at Year 3: number analyzed (Participants) | 54 | 60
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+) at Year 3 | 670.5 [319.0 to 1320.0] | 145.0 [39.0 to 349.5]
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-) at Day 0: number analyzed (Participants) | 71 | 69
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-) at Day 0 | 1.0 [1.0 to 55.0] | 1.0 [1.0 to 21.0]
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-) at Day 60: number analyzed (Participants) | 51 | 48
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-) at Day 60 | 1.0 [1.0 to 254.0] | 1.0 [1.0 to 28.0]
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-) at Year 1: number analyzed (Participants) | 84 | 79
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-) at Year 1 | 128.5 [26.0 to 281.0] | 14.0 [1.0 to 48.0]
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-) at Year 2: number analyzed (Participants) | 76 | 84
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-) at Year 2 | 1.0 [1.0 to 140.5] | 1.0 [1.0 to 34.5]
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-) at Year 3: number analyzed (Participants) | 54 | 60
  CD4.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-) at Year 3 | 244.0 [127.0 to 356.0] | 32.0 [1.0 to 77.5]
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+) at Day 0: number analyzed (Participants) | 71 | 69
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+) at Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+) at Day 60: number analyzed (Participants) | 51 | 48
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+) at Day 60 | 1.0 [1.0 to 17.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+) at Year 1: number analyzed (Participants) | 84 | 79
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+) at Year 1 | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+) at Year 2: number analyzed (Participants) | 76 | 84
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+) at Year 2 | 1.0 [1.0 to 15.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+) at Year 3: number analyzed (Participants) | 54 | 60
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+) at Year 3 | 1.5 [1.0 to 67.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-) at Day 0: number analyzed (Participants) | 71 | 69
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-) at Day 0 | 1.0 [1.0 to 23.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-) at Day 60: number analyzed (Participants) | 51 | 48
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-) at Day 60 | 1.0 [1.0 to 28.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-) at Year 1: number analyzed (Participants) | 84 | 79
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-) at Year 1 | 1.0 [1.0 to 25.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-) at Year 2: number analyzed (Participants) | 76 | 84
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-) at Year 2 | 1.0 [1.0 to 11.5] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-) at Year 3: number analyzed (Participants) | 54 | 60
  CD4.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-) at Year 3 | 1.0 [1.0 to 27.0] | 1.0 [1.0 to 6.5]
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+) at Day 0: number analyzed (Participants) | 71 | 69
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+) at Day 0 | 1.0 [1.0 to 21.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+) at Day 60: number analyzed (Participants) | 51 | 48
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+) at Day 60 | 1.0 [1.0 to 41.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+) at Year 1: number analyzed (Participants) | 84 | 79
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+) at Year 1 | 1.0 [1.0 to 28.0] | 1.0 [1.0 to 19.0]
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+) at Year 2: number analyzed (Participants) | 76 | 84
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+) at Year 2 | 1.0 [1.0 to 15.5] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+) at Year 3: number analyzed (Participants) | 54 | 60
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+) at Year 3 | 32.0 [1.0 to 107.0] | 1.0 [1.0 to 31.5]
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-) at Day 0: number analyzed (Participants) | 71 | 69
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-) at Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-) at Day 60: number analyzed (Participants) | 51 | 48
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-) at Day 60 | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-) at Year 1: number analyzed (Participants) | 84 | 79
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-) at Year 1 | 1.0 [1.0 to 19.5] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-) at Year 2: number analyzed (Participants) | 76 | 84
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-) at Year 2 | 1.0 [1.0 to 13.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-) at Year 3: number analyzed (Participants) | 54 | 60
  CD4.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-) at Year 3 | 19.0 [1.0 to 49.0] | 1.0 [1.0 to 13.0]
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+) at Day 0: number analyzed (Participants) | 71 | 69
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+) at Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 5.0]
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+) at Day 60: number analyzed (Participants) | 51 | 48
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+) at Day 60 | 1.0 [1.0 to 15.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+) at Year 1: number analyzed (Participants) | 84 | 79
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+) at Year 1 | 1.0 [1.0 to 15.0] | 1.0 [1.0 to 13.0]
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+) at Year 2: number analyzed (Participants) | 76 | 79
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+) at Year 2 | 1.0 [1.0 to 13.0] | 1.0 [1.0 to 13.0]
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+) at Year 3: number analyzed (Participants) | 54 | 60
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+) at Year 3 | 1.0 [1.0 to 24.0] | 1.0 [1.0 to 21.0]
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-) at Day 0: number analyzed (Participants) | 71 | 69
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-) at Day 0 | 1.0 [1.0 to 138.0] | 1.0 [1.0 to 114.0]
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-) at Day 60: number analyzed (Participants) | 51 | 48
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-) at Day 60 | 1.0 [1.0 to 169.0] | 25.5 [1.0 to 158.0]
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-) at Year 1: number analyzed (Participants) | 84 | 79
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-) at Year 1 | 5.0 [1.0 to 45.0] | 1.0 [1.0 to 36.0]
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-) at Year 2: number analyzed (Participants) | 76 | 84
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-) at Year 2 | 1.0 [1.0 to 30.0] | 1.0 [1.0 to 74.5]
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-) at Year 3: number analyzed (Participants) | 54 | 60
  CD4.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-) at Year 3 | 8.5 [1.0 to 128.0] | 11.0 [1.0 to 117.0]
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+) at Day 0: number analyzed (Participants) | 71 | 69
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+) at Day 0 | 74.0 [1.0 to 305.0] | 61.0 [1.0 to 181.0]
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+) at Day 60: number analyzed (Participants) | 51 | 48
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+) at Day 60 | 210.0 [48.0 to 620.0] | 91.5 [29.0 to 329.5]
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+) at Year 1: number analyzed (Participants) | 84 | 79
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+) at Year 1 | 956.0 [279.0 to 1540.5] | 159.0 [62.0 to 329.5]
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+) at Year 2: number analyzed (Participants) | 76 | 84
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+) at Year 2 | 814.5 [483.0 to 1545.5] | 215.0 [71.0 to 686.5]
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+) at Year 3: number analyzed (Participants) | 54 | 60
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+) at Year 3 | 543.5 [286.0 to 1057.0] | 112.0 [38.5 to 257.5]
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-) at Day 1: number analyzed (Participants) | 71 | 69
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-) at Day 1 | 20.0 [1.0 to 57.0] | 21.0 [1.0 to 57.0]
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-) at Day 60: number analyzed (Participants) | 51 | 48
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-) at Day 60 | 89.0 [14.0 to 185.0] | 26.0 [1.0 to 67.0]
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-) at Year 1: number analyzed (Participants) | 84 | 79
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-) at Year 1 | 152.0 [93.0 to 256.0] | 35.0 [2.0 to 98.0]
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-) at Year 2: number analyzed (Participants) | 76 | 84
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-) at Year 2 | 190.5 [95.0 to 392.0] | 52.5 [8.5 to 107.0]
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-) at Year 3: number analyzed (Participants) | 54 | 60
  CD4.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-) at Year 3 | 86.0 [45.0 to 181.0] | 25.5 [1.0 to 88.5]
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+) at Day 0: number analyzed (Participants) | 71 | 69
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+) at Day 0 | 52.0 [1.0 to 113.0] | 42.0 [9.0 to 126.0]
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+) at Day 60: number analyzed (Participants) | 51 | 48
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+) at Day 60 | 180.0 [71.0 to 422.0] | 81.0 [28.0 to 177.5]
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+) at Year 1: number analyzed (Participants) | 84 | 79
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+) at Year 1 | 41.0 [1.0 to 130.0] | 14.0 [1.0 to 39.0]
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+) at Year 2: number analyzed (Participants) | 76 | 84
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+) at Year 2 | 136.0 [49.0 to 242.0] | 22.5 [1.0 to 89.0]
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+) at Year 3: number analyzed (Participants) | 54 | 84
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+) at Year 3 | 31.0 [1.0 to 116.0] | 7.5 [1.0 to 22.0]
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-) at Day 0: number analyzed (Participants) | 71 | 69
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-) at Day 0 | 86.0 [1.0 to 184.0] | 42.0 [1.0 to 188.0]
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-) at Day 60: number analyzed (Participants) | 51 | 48
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-) at Day 60 | 242.0 [51.0 to 430.0] | 72.0 [1.0 to 186.0]
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-) at Year 1: number analyzed (Participants) | 84 | 79
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-) at Year 1 | 87.5 [39.5 to 159.5] | 9.0 [1.0 to 47.0]
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-) at Year 2: number analyzed (Participants) | 76 | 84
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-) at Year 2 | 136.5 [58.0 to 266.5] | 16.5 [1.0 to 78.5]
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-) at Year 3: number analyzed (Participants) | 54 | 60
  CD4.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-) at Year 3 | 51.5 [5.0 to 127.0] | 6.0 [1.0 to 48.5]
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+) at Day 0: number analyzed (Participants) | 71 | 69
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+) at Day 0 | 42.0 [1.0 to 124.0] | 21.0 [1.0 to 77.0]
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+) at Day 60: number analyzed (Participants) | 51 | 48
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+) at Day 60 | 186.0 [14.0 to 334.0] | 20.5 [1.0 to 118.5]
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+) at Year 1: number analyzed (Participants) | 84 | 79
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+) at Year 1 | 121.0 [28.5 to 325.5] | 28.0 [1.0 to 101.0]
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+) at Year 2: number analyzed (Participants) | 76 | 84
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+) at Year 2 | 118.0 [19.0 to 335.5] | 44.0 [1.0 to 186.0]
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+) at Year 3: number analyzed (Participants) | 54 | 60
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+) at Year 3 | 94.0 [20.0 to 267.0] | 29.0 [1.0 to 97.0]
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-) at Day 0: number analyzed (Participants) | 71 | 69
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-) at Day 0 | 1.0 [1.0 to 71.0] | 26.0 [1.0 to 99.0]
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-) at Day 60: number analyzed (Participants) | 51 | 48
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-) at Day 60 | 72.0 [1.0 to 195.0] | 16.5 [1.0 to 66.5]
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-) at Year 1: number analyzed (Participants) | 84 | 79
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-) at Year 1 | 92.5 [1.0 to 184.5] | 59.0 [1.0 to 196.0]
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-) at Year 2: number analyzed (Participants) | 76 | 84
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-) at Year 2 | 5.5 [1.0 to 124.5] | 8.5 [1.0 to 152.0]
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-) at Year 3: number analyzed (Participants) | 54 | 60
  CD4.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-) at Year 3 | 32.0 [1.0 to 190.0] | 21.0 [1.0 to 156.0]
  CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+) at Day 0: number analyzed (Participants) | 71 | 69
  CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+) at Day 0 | 71.0 [9.0 to 231.0] | 51.0 [1.0 to 128.0]
  CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+) at Day 60: number analyzed (Participants) | 51 | 48
  CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+) at Day 60 | 708.0 [158.0 to 1621.0] | 86.5 [5.0 to 381.0]
  CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+) at Year 1: number analyzed (Participants) | 84 | 79
  CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+) at Year 1 | 50.0 [7.5 to 110.0] | 22.0 [1.0 to 85.0]
  CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+) at Year 2: number analyzed (Participants) | 76 | 84
  CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+) at Year 2 | 83.0 [2.5 to 206.0] | 15.5 [1.0 to 82.0]
  CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+) at Year 3: number analyzed (Participants) | 54 | 60
  CD4.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+) at Year 3 | 35.5 [1.0 to 152.0] | 1.0 [1.0 to 45.0]

13. Secondary Outcome: Desciptive Statistics of the Frequency of M72-specific CD8+ T-cells Expressing Any Combination of Immune Markers in the Safety and Immune Sub-cohort
Description: The frequency of M72-specific CD8 + T-cells per million cells were identified after in vitro stimulation expressing any combination of immune markers ( Interleukin-2 (IL-2), cluster of differentiation 40-ligand (CD40-L), tumor necrosis factor alpha (TNF-) and interferon-gamma (IFN-) after background subtraction for each treatment group.
Time Frame: Prior to dose 1 (Day 0) and post-dose 2 (Day 60, Year 1, Year 2 and Year 3)
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: T cells per million cells
Arm/Group | M72AS01 Group | Control Group
Number analyzed (Participants) | 68 | 74
T cells per million cells
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+) at Day 0: number analyzed (Participants) | 39 | 54
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+) at Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+) at Day 60: number analyzed (Participants) | 39 | 38
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+) at Day 60 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+) at Year 1: number analyzed (Participants) | 68 | 69
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+) at Year 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+) at Year 2: number analyzed (Participants) | 67 | 74
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+) at Year 2 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+) at Year 3: number analyzed (Participants) | 42 | 53
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(+) at Year 3 | 33.5 [1.0 to 101.0] | 1.0 [1.0 to 25.0]
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-) at Day 0: number analyzed (Participants) | 56 | 54
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-) at Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-) at Day 60: number analyzed (Participants) | 39 | 38
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-) at Day 60 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-) at Year 1: number analyzed (Participants) | 68 | 69
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-) at Year 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-) at Year 2: number analyzed (Participants) | 67 | 74
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-) at Year 2 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-) at Year 3: number analyzed (Participants) | 42 | 53
  CD8.CD40L(+)+IL2(+)+TNFa(+)+IFNg(-) at Year 3 | 1.0 [1.0 to 34.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+) at Day 0: number analyzed (Participants) | 56 | 54
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+) at Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+) at Day 60: number analyzed (Participants) | 39 | 38
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+) at Day 60 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+) at Year 1: number analyzed (Participants) | 68 | 69
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+) at Year 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+) at Year 2: number analyzed (Participants) | 67 | 74
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+) at Year 2 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+) at Year 3: number analyzed (Participants) | 42 | 53
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(+) at Year 3 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-) at Day 0: number analyzed (Participants) | 56 | 54
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-) at Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-) at Day 60: number analyzed (Participants) | 39 | 38
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-) at Day 60 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-) at Year 1: number analyzed (Participants) | 68 | 69
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-) at Year 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-) at Year 2: number analyzed (Participants) | 67 | 74
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-) at Year 2 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-) at Year 3: number analyzed (Participants) | 42 | 53
  CD8.CD40L(+)+IL2(+)+TNFa(-)+IFNg(-) at Year 3 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+) at Day 0: number analyzed (Participants) | 56 | 54
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+) at Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+) at Day 60: number analyzed (Participants) | 39 | 38
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+) at Day 60 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+) at Year 1: number analyzed (Participants) | 68 | 69
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+) at Year 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+) at Year 2: number analyzed (Participants) | 67 | 74
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+) at Year 2 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+) at Year 3: number analyzed (Participants) | 42 | 53
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(+) at Year 3 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-) at Day 0: number analyzed (Participants) | 56 | 54
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-) at Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-) at Day 60: number analyzed (Participants) | 39 | 38
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-) at Day 60 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-) at Year 1: number analyzed (Participants) | 68 | 69
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-) at Year 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-) at Year 2: number analyzed (Participants) | 67 | 74
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-) at Year 2 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-) at Year 3: number analyzed (Participants) | 42 | 53
  CD8.CD40L(+)+IL2(-)+TNFa(+)+IFNg(-) at Year 3 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+) at Day 0: number analyzed (Participants) | 56 | 54
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+) at Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+) at Day 60: number analyzed (Participants) | 39 | 38
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+) at Day 60 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+) at Year 1: number analyzed (Participants) | 68 | 69
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+) at Year 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+) at Year 2: number analyzed (Participants) | 67 | 74
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+) at Year 2 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+) at Year 3: number analyzed (Participants) | 42 | 53
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(+) at Year 3 | 1.0 [1.0 to 20.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-) at Day 0: number analyzed (Participants) | 56 | 54
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-) at Day 0 | 1.0 [1.0 to 187.5] | 1.0 [1.0 to 95.0]
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-) at Day 60: number analyzed (Participants) | 39 | 38
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-) at Day 60 | 1.0 [1.0 to 112.0] | 9.5 [1.0 to 64.0]
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-) at Year 1: number analyzed (Participants) | 68 | 69
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-) at Year 1 | 1.0 [1.0 to 65.0] | 1.0 [1.0 to 41.0]
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-) at Year 2: number analyzed (Participants) | 67 | 74
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-) at Year 2 | 1.0 [1.0 to 96.0] | 4.0 [1.0 to 79.0]
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-) at Year 3: number analyzed (Participants) | 42 | 53
  CD8.CD40L(+)+IL2(-)+TNFa(-)+IFNg(-) at Year 3 | 11.5 [1.0 to 110.0] | 12.0 [1.0 to 89.0]
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+) at Day 0: number analyzed (Participants) | 56 | 54
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+) at Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+) at Day 60: number analyzed (Participants) | 39 | 38
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+) at Day 60 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+) at Year 1: number analyzed (Participants) | 68 | 69
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+) at Year 1 | 1.0 [1.0 to 43.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+) at Year 2: number analyzed (Participants) | 67 | 74
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+) at Year 2 | 45.0 [1.0 to 96.0] | 1.0 [1.0 to 37.0]
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+) at Year 3: number analyzed (Participants) | 42 | 53
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(+) at Year 3 | 42.0 [1.0 to 75.0] | 24.0 [1.0 to 51.0]
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-) at Day 0: number analyzed (Participants) | 56 | 54
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-) at Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-) at Day 60: number analyzed (Participants) | 39 | 38
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-) at Day 60 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-) at Year 1: number analyzed (Participants) | 68 | 69
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-) at Year 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-) at Year 2: number analyzed (Participants) | 67 | 74
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-) at Year 2 | 1.0 [1.0 to 27.0] | 1.0 [1.0 to 27.0]
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-) at Year 3: number analyzed (Participants) | 42 | 53
  CD8.CD40L(-)+IL2(+)+TNFa(+)+IFNg(-) at Year 3 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 14.0]
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+) at Day 0: number analyzed (Participants) | 56 | 54
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+) at Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+) at Day 60: number analyzed (Participants) | 39 | 38
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+) at Day 60 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+) at Year 1: number analyzed (Participants) | 68 | 69
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+) at Year 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+) at Year 2: number analyzed (Participants) | 67 | 74
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+) at Year 2 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+) at Year 3: number analyzed (Participants) | 42 | 53
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(+) at Year 3 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-) at Day 0: number analyzed (Participants) | 56 | 54
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-) at Day 0 | 1.0 [1.0 to 154.0] | 1.0 [1.0 to 235.0]
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-) at Day 60: number analyzed (Participants) | 39 | 38
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-) at Day 60 | 69.0 [1.0 to 225.0] | 15.5 [1.0 to 155.0]
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-) at Year 1: number analyzed (Participants) | 68 | 69
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-) at Year 1 | 1.0 [1.0 to 59.5] | 24.0 [1.0 to 73.0]
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-) at Year 2: number analyzed (Participants) | 67 | 74
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-) at Year 2 | 7.0 [1.0 to 104.0] | 1.0 [1.0 to 64.0]
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-) at Year 3: number analyzed (Participants) | 42 | 53
  CD8.CD40L(-)+IL2(+)+TNFa(-)+IFNg(-) at Year 3 | 1.0 [1.0 to 63.0] | 1.0 [1.0 to 72.0]
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+) at Day 0: number analyzed (Participants) | 56 | 54
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+) at Day 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+) at Day 60: number analyzed (Participants) | 39 | 38
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+) at Day 60 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+) at Year 1: number analyzed (Participants) | 68 | 69
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+) at Year 1 | 1.0 [1.0 to 56.5] | 1.0 [1.0 to 81.0]
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+) at Year 2: number analyzed (Participants) | 67 | 74
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+) at Year 2 | 1.0 [1.0 to 33.0] | 1.0 [1.0 to 44.0]
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+) at Year 3: number analyzed (Participants) | 42 | 53
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(+) at Year 3 | 1.0 [1.0 to 66.0] | 6.0 [1.0 to 131.0]
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-) at Day 0: number analyzed (Participants) | 56 | 54
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-) at Day 0 | 1.0 [1.0 to 22.5] | 1.0 [1.0 to 65.0]
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-) at Day 60: number analyzed (Participants) | 39 | 38
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-) at Day 60 | 19.0 [1.0 to 64.0] | 1.0 [1.0 to 2.0]
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-) at Year 1: number analyzed (Participants) | 68 | 69
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-) at Year 1 | 1.0 [1.0 to 137.5] | 1.0 [1.0 to 79.0]
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-) at Year 2: number analyzed (Participants) | 67 | 74
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-) at Year 2 | 1.0 [1.0 to 156.0] | 1.0 [1.0 to 125.0]
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-) at Year 3: number analyzed (Participants) | 42 | 53
  CD8.CD40L(-)+IL2(-)+TNFa(+)+IFNg(-) at Year 3 | 1.0 [1.0 to 104.0] | 1.0 [1.0 to 313.0]
  CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+) at Day 0: number analyzed (Participants) | 56 | 54
  CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+) at Day 0 | 26.0 [1.0 to 750] | 13.5 [1.0 to 2701]
  CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+) at Day 60: number analyzed (Participants) | 39 | 38
  CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+) at Day 60 | 18.0 [1.0 to 477] | 1.0 [1.0 to 1033]
  CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+) at Year 1: number analyzed (Participants) | 68 | 69
  CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+) at Year 1 | 1.5 [1.0 to 2981] | 1.0 [1.0 to 2819]
  CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+) at Year 2: number analyzed (Participants) | 67 | 74
  CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+) at Year 2 | 1.0 [1.0 to 978] | 3.0 [1.0 to 777]
  CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+) at Year 3: number analyzed (Participants) | 42 | 53
  CD8.CD40L(-)+IL2(-)+TNFa(-)+IFNg(+) at Year 3 | 1.0 [1.0 to 1384] | 16.0 [1.0 to 537]

14. Secondary Outcome: M72-specific Antibody Concentrations as Measured by Enzyme Linked Immuno Sorbent Assay (ELISA) in the Safety and Immune Sub-cohort
Description: Mycobacterium tuberculosis M72-specific antibody geometric mean concentrations (GMCs) with exact 95% Confidence Interval (CI) were measured by Enzyme Linked Immuno Sorbent Assay (ELISA) and expressed in ELISA unit per milliliter (EU/mL). The cut-off of the assay was 2.8 EU/mL. The Geometric Mean Concentration (GMC) calculations were performed by taking the anti-log of the mean of the log10 concentration transformations. For descriptive statistics purposes only, antibody concentrations below the cut-off value of the assay was given an arbitrary value of half the cut-off value for the purpose of GMC calculation.
Time Frame: Prior to dose 1 (Day 0) and post-dose 2 (Day 60, Year 1, Year 2 and Year 3)
Population: Analysis was performed on the "safety and immunogenicity" sub-cohort (i.e. about 150 subjects enrolled in each group and from 2 of the 3 countries [the third country study start was delayed as awaiting regulatory approval]) which included subjects with at least 1 cell-mediated immune result documented.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | M72AS01 Group | Control Group
Number analyzed (Participants) | 120 | 124
EU/mL
  Anti-M72 at Day 0 | 1.6 [1.5 to 1.8] | 1.6 [1.5 to 1.7]
  Anti-M72 at Day 60: number analyzed (Participants) | 99 | 97
  Anti-M72 at Day 60 | 547.0 [471.1 to 635.1] | 1.6 [1.4 to 1.7]
  Anti-M72 at Year 1: number analyzed (Participants) | 118 | 119
  Anti-M72 at Year 1 | 41.5 [35.4 to 48.6] | 1.7 [1.5 to 1.8]
  Anti-M72 at Year 2: number analyzed (Participants) | 108 | 114
  Anti-M72 at Year 2 | 30.6 [26.2 to 35.6] | 1.6 [1.5 to 1.8]
  Anti-M72 at Year 3: number analyzed (Participants) | 83 | 92
  Anti-M72 at Year 3 | 27.0 [22.7 to 32.0] | 1.6 [1.4 to 1.7]

15. Secondary Outcome: Number of Seropositive Subjects for M72 Antibodies Measured by ELISA in the Safety and Immune Sub-cohort
Description: A seronegative subject was a subject whose antibody concentration was below 2.8 EU/mL, while a seropositive subject was a subject whose antibody concentration was greater than or equal to 2.8 EU/mL.
Time Frame: Prior to dose 1 (Day 0) and post-dose 2 (Day 60, Year 1, Year 2 and Year 3)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | M72AS01 Group | Control Group
Number analyzed (Participants) | 120 | 124
Participants
  Anti-M72 at Day 0 | 11 | 12
  Anti-M72 at Day 60: number analyzed (Participants) | 99 | 97
  Anti-M72 at Day 60 | 99 | 8
  Anti-M72 at Year 1: number analyzed (Participants) | 118 | 119
  Anti-M72 at Year 1 | 117 | 14
  Anti-M72 at Year 2: number analyzed (Participants) | 108 | 114
  Anti-M72 at Year 2 | 108 | 11
  Anti-M72 at Year 3: number analyzed (Participants) | 83 | 92
  Anti-M72 at Year 3 | 83 | 8

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms were reported during the 7-day (Days 0-6) post-vaccination period and unsolicited AE(s): during the 30-day (Days 0-29) post-vaccination period. SAE(s): were reported during the entire study period (from Month 0 to Month 36 (Year 3).
Arm/Group | M72AS01 Group | Control Group
All-Cause Mortality (participants affected / at risk) | 19/1786 | 28/1787
Serious Adverse Events (participants affected / at risk) | 51/1786 | 62/1787
Other Adverse Events (participants affected / at risk) | 1204/1786 | 809/1787
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | M72AS01 Group (N=1786) | Control Group (N=1787)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Basedow's disease (Endocrine disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Accidental death (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 3 (3) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Acute hiv infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2)
Lymph node tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Malaria (Infections and infestations) | 2 (2) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 2 (3) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis gastrointestinal (Infections and infestations) | 0 (0) | 1 (1)
Typhoid fever (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Crush injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 4 (4) | 11 (11)
Head injury (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stab wound (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Schizophrenia (Psychiatric disorders) | 0 (0) | 1 (1)
Substance abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Substance-induced psychotic disorder (Psychiatric disorders) | 2 (2) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | M72AS01 Group (N=1786) | Control Group (N=1787)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 3 (3)
Eosinophilia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Lymph node calcification (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 13 (15) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Ear disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 4 (4) | 6 (6)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Motion sickness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 3 (3) | 6 (6)
Eye discharge (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 11 (11) | 5 (6)
Eye pruritus (Eye disorders) | 2 (2) | 3 (4)
Eye swelling (Eye disorders) | 4 (4) | 2 (2)
Eyelid cyst (Eye disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 4 (4) | 3 (3)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 5 (5) | 6 (7)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 59 (64) | 48 (61)
Abdominal pain lower (Gastrointestinal disorders) | 3 (3) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 23 (28) | 28 (30)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3) | 3 (3)
Dental caries (Gastrointestinal disorders) | 4 (4) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 45 (50) | 30 (37)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 5 (6)
Enteritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric disorder (Gastrointestinal disorders) | 5 (5) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 8 (8) | 9 (11)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 3 (3)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 3 (4)
Lip blister (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 47 (52) | 25 (26)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral contusion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 3 (3)
Proctalgia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 16 (19) | 22 (25)
Vomiting (Gastrointestinal disorders) | 34 (35) | 16 (16)
Administration site pain (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 19 (22) | 7 (8)
Axillary pain (General disorders) | 4 (4) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 30 (31) | 19 (22)
Chills (General disorders) | 72 (78) | 8 (9)
Facial pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 115 (134) | 51 (58)
Feeling cold (General disorders) | 12 (12) | 5 (5)
Feeling hot (General disorders) | 33 (38) | 17 (20)
Feeling of body temperature change (General disorders) | 1 (1) | 0 (0)
Hangover (General disorders) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 1 (3) | 1 (1)
Ill-defined disorder (General disorders) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 14 (14) | 11 (11)
Injection site bruising (General disorders) | 1 (1) | 1 (1)
Injection site discolouration (General disorders) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 65 (66) | 1 (1)
Injection site hypersensitivity (General disorders) | 1 (1) | 0 (0)
Injection site hypoaesthesia (General disorders) | 3 (3) | 0 (0)
Injection site induration (General disorders) | 4 (4) | 0 (0)
Injection site joint pain (General disorders) | 4 (4) | 0 (0)
Injection site lymphadenopathy (General disorders) | 2 (2) | 0 (0)
Injection site movement impairment (General disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 616 (848) | 75 (87)
Injection site papule (General disorders) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 27 (29) | 5 (6)
Injection site rash (General disorders) | 9 (9) | 1 (1)
Injection site reaction (General disorders) | 13 (15) | 1 (1)
Injection site swelling (General disorders) | 192 (221) | 7 (7)
Injection site vesicles (General disorders) | 1 (1) | 0 (0)
Injection site warmth (General disorders) | 0 (0) | 1 (1)
Injury associated with device (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 35 (35) | 5 (6)
Pain (General disorders) | 63 (74) | 10 (11)
Peripheral swelling (General disorders) | 5 (6) | 2 (2)
Pyrexia (General disorders) | 121 (142) | 22 (22)
Suprapubic pain (General disorders) | 1 (1) | 0 (0)
Swelling (General disorders) | 0 (0) | 2 (2)
Thirst (General disorders) | 1 (1) | 0 (0)
Vaccination site pain (General disorders) | 1 (1) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 6 (6)
Vessel puncture site pruritus (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 1 (1)
Food allergy (Immune system disorders) | 0 (0) | 2 (2)
Hypersensitivity (Immune system disorders) | 2 (3) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 3 (3)
Abscess jaw (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 2 (2) | 2 (2)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1)
Amoebiasis (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Anorectal infection (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Ascariasis (Infections and infestations) | 1 (1) | 0 (0)
Atypical mycobacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 1 (1) | 0 (0)
Body tinea (Infections and infestations) | 2 (2) | 2 (2)
Breast abscess (Infections and infestations) | 0 (0) | 1 (2)
Bronchitis (Infections and infestations) | 1 (1) | 3 (3)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Carbuncle (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 3 (3) | 2 (2)
Cervicitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 5 (5) | 6 (6)
Conjunctivitis bacterial (Infections and infestations) | 3 (3) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Dysentery (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 3 (3) | 4 (4)
Fungal skin infection (Infections and infestations) | 3 (3) | 3 (3)
Furuncle (Infections and infestations) | 0 (0) | 3 (3)
Gastroenteritis (Infections and infestations) | 7 (7) | 16 (16)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Gingival abscess (Infections and infestations) | 0 (0) | 2 (2)
Gingivitis (Infections and infestations) | 0 (0) | 2 (2)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 2 (2)
Helminthic infection (Infections and infestations) | 2 (2) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 2 (2)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Hiv infection (Infections and infestations) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 1 (1) | 0 (0)
Infected bite (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 62 (67) | 51 (54)
Injection site abscess (Infections and infestations) | 1 (1) | 0 (0)
Injection site pustule (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 5 (5) | 8 (8)
Malaria (Infections and infestations) | 52 (53) | 54 (57)
Nasopharyngitis (Infections and infestations) | 14 (14) | 15 (15)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 4 (4)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 4 (4)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 1 (1) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 9 (10) | 10 (10)
Pneumonia (Infections and infestations) | 2 (2) | 3 (4)
Rash pustular (Infections and infestations) | 2 (2) | 1 (1)
Respiratory tract infection (Infections and infestations) | 4 (4) | 7 (7)
Rhinitis (Infections and infestations) | 22 (24) | 29 (29)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sexually transmitted disease (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 6 (6) | 8 (9)
Skin bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 4 (4) | 1 (2)
Tinea capitis (Infections and infestations) | 1 (1) | 0 (0)
Tinea infection (Infections and infestations) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 2 (2)
Tinea versicolour (Infections and infestations) | 5 (5) | 4 (4)
Tonsillitis (Infections and infestations) | 4 (4) | 7 (7)
Tooth abscess (Infections and infestations) | 2 (2) | 3 (3)
Typhoid fever (Infections and infestations) | 3 (3) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 64 (70) | 72 (76)
Urethritis (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 9 (10) | 15 (16)
Vaginal infection (Infections and infestations) | 0 (0) | 3 (3)
Varicella (Infections and infestations) | 0 (0) | 3 (3)
Viral rash (Infections and infestations) | 0 (0) | 1 (1)
Vulval abscess (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 3 (3) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 2 (3)
Wound infection (Infections and infestations) | 2 (2) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Animal bite (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Heat stroke (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injection related reaction (Injury, poisoning and procedural complications) | 1 (2) | 1 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 3 (4) | 3 (3)
Limb injury (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Penis injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Scar (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 4 (4) | 8 (8)
Soft tissue injury (Injury, poisoning and procedural complications) | 6 (6) | 3 (3)
Stab wound (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 2 (6) | 3 (3)
Wound (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Alanine aminotransferase increased (Investigations) | 4 (4) | 6 (6)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 5 (5)
Blood pressure diastolic increased (Investigations) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 5 (5) | 4 (4)
Blood pressure systolic increased (Investigations) | 3 (3) | 3 (3)
Body temperature decreased (Investigations) | 0 (0) | 1 (3)
Body temperature increased (Investigations) | 2 (2) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 6 (6) | 3 (3)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Hiv test positive (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 9 (9) | 6 (6)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (2) | 0 (0)
Respiratory rate increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 12 (12) | 8 (8)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1)
White blood cell count increased (Investigations) | 2 (2) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 33 (34) | 11 (11)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminanemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 (31) | 21 (22)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Arthropathy (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 66 (76) | 32 (35)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (8)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 (11) | 10 (11)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 84 (88) | 25 (28)
Myositis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 15 (17) | 6 (7)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 26 (30) | 18 (18)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 120 (132) | 93 (104)
Headache (Nervous system disorders) | 620 (879) | 341 (483)
Hypoaesthesia (Nervous system disorders) | 7 (7) | 4 (4)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 2 (2)
Neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Optic neuritis (Nervous system disorders) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 3 (3) | 1 (1)
Poor quality sleep (Nervous system disorders) | 1 (1) | 0 (0)
Post-traumatic headache (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 5 (5) | 3 (3)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Tension headache (Nervous system disorders) | 2 (2) | 6 (6)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 4 (4)
Libido increased (Psychiatric disorders) | 2 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Micturition disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral discharge (Renal and urinary disorders) | 1 (1) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 6 (6) | 7 (7)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Genital ulceration (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 4 (4) | 6 (6)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Penile discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pruritus genital (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Scrotal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 32 (33) | 38 (39)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (6)
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 15 (16)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 10 (10)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (6)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 12 (12) | 4 (4)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 13 (15) | 3 (3)
Penile ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 8 (8) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 16 (19) | 18 (18)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Trichorrhexis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Bloody discharge (Vascular disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 6 (6) | 5 (5)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 2 (2)
Systolic hypertension (Vascular disorders) | 2 (2) | 0 (0)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Vascular pain (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2014-01-29): https://cdn.clinicaltrials.gov/large-docs/98/NCT01755598/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-17): https://cdn.clinicaltrials.gov/large-docs/98/NCT01755598/SAP_001.pdf